CLINICAL TRIAL: NCT06443255
Title: Comparison of Cocaine, Lidocaine/xylometazoline and Saline for Intranasal Analgesia - a Blinded Triple Crossover Study
Brief Title: Cocaine, Lidocaine/xylometazoline and Saline for Nasal Analgesia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Mo Haslund Larsen, Principal investigator, Rigshospitalet, Denmark
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2023-506644-17
Record Dates: First submitted 2024-05-29; First posted 2024-06-05 (Actual); Last update posted 2024-09-27 (Actual); Status verified 2024-07

CONDITIONS: Analgesia
MeSH Terms: conditions — Agnosia | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Cocaine (Active Comparator): 2 mL 4% cocaine hydrochloride
  Interventions: Drug: Cociane hydrochloride 4%
- Xylometazoline and lidocaine (Active Comparator): 1.5 mL of 4% lidocaine and 0.5 mL 0.1% xylometazoline
  Interventions: Drug: Lidocaine 4%; Drug: Xylometazoline 0.1%
- Saline (Placebo Comparator): 2 ml of 0,9% saline solution
  Interventions: Drug: Saline 0.9%

INTERVENTIONS:
Drug: Cociane hydrochloride 4% — 2 mL of 4% cocaine
  Arms: Cocaine
Drug: Lidocaine 4% — 1.5 mL of 4% lidocaine
  Arms: Xylometazoline and lidocaine
Drug: Xylometazoline 0.1% — 0.5 mL of xylometazoline 0.1%
  Arms: Xylometazoline and lidocaine
Drug: Saline 0.9% — 2 mL of saline 0.9%
  Arms: Saline

SUMMARY:
When performed by trained personnel nasotracheal intubation is a safe and effective technique for attaining a secure airway in preparation for surgery of the head and neck. The procedure can be deemed necessary due to the nature of the surgical procedure or considerations in regard to the patient's comorbidities. For a certain group of patients with expected difficult airways, the procedure is done whilst they are awake and aided by fiberoptics.

For these awake patients, extra precautions must be taken to ensure the procedure is conducted with minimal pain and discomfort. The pain and discomfort arises from the mechanical manipulation of the nasal mucosa and can be alleviated in part by means of topical analgesia as well as through decongestion, providing more space within the nasal cavity. For these purposes, several drugs in varying combinations and dosages are used, but no single drug choice is universally recommended.

Cocaine is one of these appropriate drugs. It is a magistral formula used especially due to its unique combination of both vasoconstrictive and analgesic properties. Concerns have though been raised regarding cocaine's potential toxicity and alternative medications are continuously sought after.

A combination of lidocaine and xylometazoline can also be used for preparation of the nose prior to awake nasal fiberoptic intubation. Lidocaine contributes with its analgesic effect whilst xylometazoline functions as the vasoconstrictor.

The investigators wish to compare the analgesic effects of cocaine and lidocaine/phenylephrine to each other and saline when subjectively scored on a visual analogue scale of 0-100 mm immediately after simulated awake nasal intubation on healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Proficient in spoken and written Danish
* Healthy volunteers (no active diagnoses)
* Negative hCG (human chorionic gonadotropin) urine stix for women of childbearing potential

Exclusion Criteria:

* Known nasal malformation
* Known coagulopathy
* Current antithrombotic treatment
* Self-reported epistaxis occurring more than once a month
* Symptoms of a common cold within the past week
* Hypersensitivity to local anaesthetics of amide type or any of the excipients
* Hypertension
* Narrow-angle glaucoma

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2024-07-01 (Actual); Primary Completion 2024-08-27 (Actual); Study Completion 2024-08-27 (Actual)

PRIMARY OUTCOMES:
Pain regarding the procedure | Immediately following the procedure of 10 cm insertion of a 6.0 nasal endotracheal tube
  Self reported pain on a visual analogue scale of 0-100 mm

SECONDARY OUTCOMES:
Pain regarding the procedure | One minute after the procedure of insertion of a 6.0 nasal endotracheal tube
  Self reported pain on a visual analogue scale of 0-100 mm
Volume | 5 minutes before drug administration and 1, 3, 5, 7 and 9 minutes after drug administration
  Volume within both nasal cavities measured with acoustic rhinometry
Fiberoptic endoscopy | Fiberoptic endoscopy performed 10 minutes before drug administraion and 10 minutes after drug administration
  Preferred nasal cavity based on a comparison of the degree of vasoconstriction of the nasal mucosa evaluated by fiberoptic endoscopy assessed by ENT-specialist
Drug test detection | 15 minutes before drug administration and 1, 2 and 3 hours after drug administration
  Concentraion of cocaine and cocaine's main metabolite benzoylecgonine in blood and saliva samples respectively
Heart rate | 5 minutes before drug administration and 1, 2, 3, 4 and 5 minutes after drug administration
  Measurement of heart rate
Blood pressure | 5 minutes before drug administration and 1, 2, 3, 4 and 5 minutes after drug administration
  Measurement of mean arterial blood pressure
Patient-centred questions | 15 minutes after drug administration
  The degree of discomfort and unpleasentness of taste of the drug administration on a scale of 1-10 and whether they felt exaltation after drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Mo H Larsen, MD, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Rigshospitalet, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Larsen MH, Rosenkrantz O, Knudsen RL, Hesselfeldt R, Hilberg O, Siersma V, Heiberg J, Rasmussen LS, Isbye D. Analgesic Effect of Cocaine and Lidocaine/Xylometazoline in Healthy Volunteers Undergoing Awake Nasal Intubation: A Randomized Controlled Crossover Trial. Acta Anaesthesiol Scand. 2025 Jul;69(6):e70056. doi: 10.1111/aas.70056. PMID 40346884